CLINICAL TRIAL: NCT04413734
Title: Combination of Anti-PD-1 Antibody and Chemotherapy for Unresectable Intrahepatic Cholangiocarcinoma: A Exploratory Clinical Trial
Brief Title: Combination of Anti-PD-1 Antibody and Chemotherapy for Unresectable Intrahepatic Cholangiocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Clinical Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CISLD-9
Record Dates: First submitted 2020-05-30; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Intrahepatic Cholangiocarcinoma by AJCC V8 Stage
Keywords: Intrahepatic Cholangiocarcinoma; Immunotherapy; anti-programmed-death-1 antibody
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Combined Modality Therapy; Immunotherapy; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triprilumab in combination with chemotherapy of GP (Experimental): Triprilumab, 240 mg, every 3 weeks (Q3W), Day 1 of each 3 week cycle PLUS Gemcitabine, 1000 mg/m^2, Q3W, Day 1 and Day 8 of each cycle PLUS Cisplatin, 25 mg/m^2, Q3W, Day 1 and Day 8 of each cycle until progressive disease or unacceptable toxicity .
  Interventions: Drug: Combination therapy
- Mono-chemotherapy of GP (Active Comparator): Gemcitabine, 1000 mg/m^2, Q3W, Day 1 and Day 8 of each cycle PLUS Cisplatin, 25 mg/m^2, Q3W, Day 1 and Day 8 of each cycle until progressive disease or unacceptable toxicity.
  Interventions: Drug: Mono-chemotherapy

INTERVENTIONS:
Drug: Combination therapy — Triprilumab by intravenous infusion accompanying with Gemcitabine plus Cisplatin
  Other Names: Triprilumab; Immunotherapy; Anti-PD-1 therapy
  Arms: Triprilumab in combination with chemotherapy of GP
Drug: Mono-chemotherapy — Gemcitabine plus Cisplatin by intravenous infusion
  Other Names: Gemcitabine Injection plus Cisplatin Injection
  Arms: Mono-chemotherapy of GP

SUMMARY:
This study is designed to observe and evaluate the safety and the efficacy of the anti-programmed-death-1 antibody (anti-PD-1) Triprilumab in combination with chemotherapy of Gemcitabine PLUS Cisplatin in patients who were advanced intrahepatic cholangiocarcinoma with no chance for primary surgery.

DETAILED DESCRIPTION:
Intrahepatic cholangiocarcinoma, also known as intrahepatic cholangiocarcinoma, is derived from intrahepatic bile duct epithelial cells, the second most common primary liver malignant tumor in china. but most (60% -70%) patients is diagnosed at the advanced stage . Gemcitabine plus cisplatin is the standard first-line advanced treatment recommended in international and domestic guidelines, but the treatment effect remains to be improved.

The clinical benefits of immune therapies for HCC are emerging. Early clinical data already show the safety of immune checkpoint inhibition. This study is to analyze the safety and efficacy of immunotherapy Triprilumab Injection combined with Gemcitabine Injection plus Cisplatin Injection in patients with advanced intrahepatic cholangiocarcinoma.

Patients who were aged 18 to 80 years with a histological or cytological diagnosis of intrahepatic cholangiocarcinoma，locally advanced or multiple liver metastases, including postoperative occurrence, will be enrolled in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically confirmed diagnosis of advanced (metastatic) and/or unresectable (locally advanced) biliary tract cancer (intra-or extrahepatic cholangiocarcinoma)
* Has at least one measurable, evaluable lesions based on Response Evaluation Criteria in Solid Tumors (RECIST 1.1), as determined by the research center investigator
* Participants with a history of hepatitis B or hepatitis C can be enrolled if they meet study criteria
* Is willing to provide archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion
* Has a life expectancy of greater than 3 months
* Has adequate organ function
* Has EOCG score 0 or 1
* Has willing to voluntarily participate in clinical trial and sign informed consent

Exclusion Criteria:

* Histology includes fibrolamellar, hepatocytes, sarcomatoid liver cancer, hepatocytes, hepatocellular carcinoma and other components. Or has had previous biliary tract cancer (intra-or extra hepatic cholangiocarcinoma) or combined with other cancer with an exception of basal cell carcinoma and squamous cell carcinoma of the skin carcinoma in situ that has been radical treated.
* Has active tuberculosis and were receiving anti-tb treatment, or receiving anti-tb treatment within a year before were randomly assigned.
* Has symptomatic or poorly controlled circulatory disease, such as Congestive heart failure(NYHA III-IV), arrhythmia instability, type I angina, coronary heart disease, etc
* Has esophageal and gastric varices bleeding due to portal hypertension, or with history of inflammatory bowel disease, gastrointestinal perforation and intestinal obstruction, abdominal abscess, or chronic diarrhea.
* Has life-threatening bleeding or venous thromboembolism events occurred in the first six months before enrollment, or the patient was prone to severe bleeding or coagulation dysfunction, or was undergoing thrombolytic therapy
* Has active autoimmune disease requiring systemic treatment within the two years before enrollment , especially those with immunosuppressive drugs, who were unable to control or who needed large amounts of immunosuppressive drugs to control the disease, excluding topical glucose-corticosteroids or systemic use, and prednisone less than 10 milligrams per day
* Has central nervous system disease with symptoms, such as primary brain tumor, stroke, epilepsy, etc. Patients who have undergone central nervous system or known brain metastases
* Has acute or severe hepatitis infection, or a severe bacterial or bacterial infection in an active or clinically poorly controlled, or with congenital or acquired immune deficiency such human immunodeficiency virus (HIV) infected
* Has previous allogeneic stem cell or parenchymal organ transplantation, including after liver transplantation
* Has history of allergies to drugs involved in this study
* Women who are pregnant or lactating, or who do not want to use contraception during the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-04-22 (Actual); Primary Completion 2022-04-22 (Estimated); Study Completion 2024-04-22 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Observation period 48 months
  Time from first randomization to the first documented disease progression or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 48 months
  Overall survival is defined as the time from randomization to death due to any cause.
Objective Response Rate (ORR) per RECIST 1.1 | Up to 48 months
  ORR is defined as the percentage of participants who have a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: a ≥30% decrease in the sum of diameters [SOD] of target lesions) as assessed by RECIST 1.1
Disease Control Rate(DCR) | Up to 48 months
  DCR is defined as the percentage of participants who have a confirmed Complete Response or Partial Response as assessed by RECIST 1.1
Myopathologic response(MPR) | Up to 48 months
  DCR is defined as the proportion of patients with residual survival tumor ≤10%, the evaluation requires two liver cancer pathologists to evaluate and judge. If the difference between the two pathologists' evaluation is ≤10%, the average value is taken as the pathological remission rate. If the difference is greater than 10%, a third pathologist is required to evaluate, and then the average of the two with a difference of less than 10% will be taken
Conversion surgical resection(R0) rate | Up to 48 months
  the ratio of patients successfully converted into radical surgical resection by the treatment plan, in which the margin of the liver is negative
Adverse Events (AE) | Up to 48 months
  Safety evaluation was done continuously during treatment by using CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China